CLINICAL TRIAL: NCT00005981
Title: Phase II Trial of O6Benzylguanine and BCNU in Patients With Colon and Rectal Carcinoma
Brief Title: Combination Chemotherapy in Treating Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Smitha Krishnamurthi, MD, Ireland Cancer Center at University Hospitals Cancer Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU1298; U01CA063200 (NIH); P30CA043703 (NIH); CWRU-1298; NCI-89
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2010-06

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — O(6)-benzylguanine; Carmustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: O6-benzylguanine — Patients receive O6-benzylguanine (BG) IV over 1 hour. Treatment continues every 6 weeks in the absence of disease progression or unacceptable toxicity.
Drug: carmustine — Carmustine IV over 1 hour (beginning 1 hour after completion of BG infusion) on day 1. Treatment continues every 6 weeks in the absence of disease progression or unacceptable toxicity.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients who have metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate of patients with metastatic colorectal carcinoma treated with O6-benzylguanine and carmustine.
* Evaluate tumor tissue biochemical and immunohistochemical predictors of response in patients treated with this regimen.
* Correlate carcinoembryonic antigen levels in the peripheral blood with response in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive O6-benzylguanine (BG) IV over 1 hour and carmustine IV over 1 hour (beginning 1 hour after completion of BG infusion) on day 1. Treatment continues every 6 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 19-36 patients will be accrued for this study within 1.7-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of metastatic colorectal carcinoma
* Bidimensionally measurable disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* WBC at least 4,000/mm^3
* Granulocyte count at least 1,500/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin greater than 8 g/dL

Hepatic:

* Bilirubin no greater than 1.2 mg/dL
* AST and ALT less than 2.5 times upper limit of normal (ULN)
* PT no greater than ULN (not on anticoagulation therapy)

Renal:

* Creatinine no greater than 1.5 mg/dL
* Creatine clearance greater than 60 mL/min

Pulmonary:

* DLCO at least 60%

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after study
* No other concurrent active malignancies
* Prior malignancies presumed to be cured allowed
* No other concurrent uncontrolled severe medical problem that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 6 months since prior adjuvant chemotherapy without disease recurrence
* No more than 1 prior chemotherapy regimen for metastatic disease

Endocrine therapy:

* Not specified

Radiotherapy:

* Prior adjuvant radiotherapy allowed
* No prior radiotherapy to more than 25% of total bone marrow

Surgery:

* Not specified

Other:

* No other prior therapy for advanced disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2000-06; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Determine the response rate of patients with metastatic colorectal carcinoma treated with O6-benzylguanine and carmustine. | Treatment continues every 6 weeks in the absence of disease progression or unacceptable toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Smitha Krishnamurthi, MD, Study Chair — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States